CLINICAL TRIAL: NCT01383616
Title: Unipedicular vs. Bipedicular Kyphoplasty for the Treatment of Osteoporotic Vertebral Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 26033
Record Dates: First submitted 2011-06-13; First posted 2011-06-28 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Vertebral Compression Fracture
Keywords: osteoporosis; vertebral compression fractures
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unipedicular kyphoplasty (Active Comparator): Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm only vertebral body pedicle was entered to deliver bone cement.
  Interventions: Device: Kyphon® Balloon Kyphoplasty (Kyphon Inc; Sunnydale, CA)
- Bipedicular Kyphoplasty group (Active Comparator): Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm two pedicles were entered to deliver bone cement.
  Interventions: Device: Kyphon® Balloon Kyphoplasty (Kyphon Inc; Sunnydale, CA)

INTERVENTIONS:
Device: Kyphon® Balloon Kyphoplasty (Kyphon Inc; Sunnydale, CA) — A Jamshidi Crown Bone Biopsy Needle (Cardinal Health; Dublin, OH) was then introduced through the incision into the pedicle, and advanced through the pedicle into the center of the vertebral body using a mallet at a 30 to 45 degree angle relative to the AP axis. A guidewire was then placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated until the balloon was in contact with the subchondral plate, lateral vertebral body wall, or anterior cortex of the vertebral body. The balloon was then deflated and removed. Subsequently, cement was injected into the cavity and allowed to harden.

SUMMARY:
Balloon kyphoplasty for the treatment of patients with osteoporotic vertebral compression fractures has been shown to be successful in providing acute pain relief, enabling improved function, and restoring of vertebral body height. However, limited prospective data exists in the investigation of unipedicular balloon kyphoplasty as a sufficient alternative to bipedicular balloon kyphoplasty. The purpose of this prospective randomized study was to compare the clinical and radiographic outcomes of unipedicular and bipedicular balloon kyphoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Males or females older than 50 years of age with acute vertebral compression fractures causing significant pain and functional limitations in their daily activities.

Exclusion Criteria:

* primary tumors of bone or evidence of metastasis at the index vertebrae
* pre-existing chronic pain or functional disability unrelated to a vertebral compression fracture which would confound the data analysis
* fracture secondary to a traumatic event
* inability to fully visualize both pedicles of the fractured vertebrae on intraoperative fluoroscopy

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tzipora Kuba, PhD, Study Director — Hospital for Special Surgery, New York; Joseph M Lane, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Unipedicular Kyphoplasty: Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm only vertebral body pedicle was entered to deliver bone cement. Kyphon® Balloon Kyphoplasty (Kyphon Inc; Sunnydale, CA): A Jamshidi Crown Bone Biopsy Needle (Cardinal Health; Dublin, OH) was then introduced through the incision into the pedicle, and advanced through the pedicle into the center of the vertebral body using a mallet at a 30 to 45 degree angle relative to the AP axis. A guidewire was then placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated.
- Bipedicular Kyphoplasty Group: Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm two pedicles were entered to deliver bone cement. Kyphon® Balloon Kyphoplasty (Kyphon Inc; Sunnydale, CA): A Jamshidi Crown Bone Biopsy Needle (Cardinal Health; Dublin, OH) was then introduced through the incision into the pedicle, and advanced through the pedicle into the center of the vertebral body using a mallet at a 30 to 45 degree angle relative to the AP axis. A guidewire was then placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated.
Period: Overall Study
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Started | 40 | 44
Completed | 23 | 21
Not Completed | 17 | 23

BASELINE CHARACTERISTICS:
Population: 21 patients received bipedicular intervention. 3 lost to follow up at 3 months (n=18) and 6 total lost at 12 months (n=15) 23 patients received unipedicular intervention. 5 lost to 3 month follow up (n=18) and 9 total lost at 12 months (n=14) Pre and post-op vertebral height measures were available in 14 unipedicular and 17 bipedicular patients
Groups:
- Unipedicular Kyphoplasty: In this arm only vertebral body pedicle was entered to deliver bone cement. Kyphon® Balloon Kyphoplasty (Kyphon Inc; Sunnydale, CA): A Jamshidi Crown Bone Biopsy Needle (Cardinal Health; Dublin, OH) was then introduced through the incision into the pedicle, and advanced through the pedicle into the center of the vertebral body using a mallet at a 30 to 45 degree angle relative to the AP axis. A guidewire was then placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated until the balloon was in contact with the subchondral plate, lateral vertebral body wall, or anterior cortex of the vertebral body. The balloon was then deflated and removed. Subsequently, cement was injected into the cavity and allowed to harden.
- Bipedicular Kyphoplasty Group: In this arm two pedicles were entered to deliver bone cement. Kyphon® Balloon Kyphoplasty (Kyphon Inc; Sunnydale, CA): A Jamshidi Crown Bone Biopsy Needle (Cardinal Health; Dublin, OH) was then introduced through the incision into the pedicle, and advanced through the pedicle into the center of the vertebral body using a mallet at a 30 to 45 degree angle relative to the AP axis. A guidewire was then placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated until the balloon was in contact with the subchondral plate, lateral vertebral body wall, or anterior cortex of the vertebral body. The balloon was then deflated and removed. Subsequently, cement was injected into the cavity and allowed to harden.
- Total: Total of all reporting groups
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 23 | 21 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.7 (7.8) | 79.3 (6.5) | 79 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Comparison of 3 Month ODI Score Between Unipedicular and Bipedicular Kyphoplasty Groups
Description: The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. The self-completed questionnaire contains ten topics. Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Time Frame: Preoperative questionnaire within 3 weeks before surgery and postoperative questionnaires at 3 months after surgery
Population: From the period of intervention to 3 month follow-up, 5 patients were lost in the unipedicular kyphoplasty arm, resulting in analysis of 18 patients from this arm at 3 months. 3 patients were lost in the bipedicular kyphoplasty arm, resulting in analysis of 18 patients from this arm at 3 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 18 | 18
units on a scale | 15 (4) | 14 (5)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Comparison of 3 month ODI Score between Unipedicular and Bipedicular kyphoplasty groups; Test type: Superiority; p = 0.85, t-test, 2 sided

2. Primary Outcome: Change in RDQ in the Bipedicular Group From 3 to 12 Months
Description: The Roland Morris Disability Questionnaire is a widely used health status measure for low back pain. The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore vary from 0 to 24. It is not recommended to give patients a 'Yes' / 'No' option. If patients indicate in any way that an item is not applicable to them, the item is scored 'No', i.e. the denominator remains 24. A score of 0 indicates no low back pain, while a score of 24 indicates significant low back pain.
Time Frame: 3-12 months post operation
Population: From the period of intervention to 12 month follow-up, 6 total patients were lost in the bipedicular kyphoplasty arm, resulting in analysis of 15 patients from this arm at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bipedicular Kyphoplasty Group: Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm two pedicles were entered deliver bone cement.
  A guidewire was placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated until the balloon was in contact with the subchondral plate, lateral vertebral body wall, or anterior cortex of the vertebral body. The balloon was then deflated and removed. Subsequently, cement was injected into the cavity and allowed to harden.
Arm/Group | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 15
units on a scale | 4.7 (1.8)
Statistical Analysis 1: Comparison: Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.008, t-test, 2 sided

3. Secondary Outcome: Anterior Vertebral Body Height Restoration Following Surgery With Kyphoplasty
Description: Preoperative and postoperative thoracolumbar radiographs were used to calculate the percent changes of the anterior vertebral body heights.
Time Frame: Preoperative assessment within 3 weeks before surgery and postoperative day 1
Population: Pre and postoperative measurements were available for 14 patients in the unipedicular group, and 17 patients in the bipedicular group.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 14 | 17
percent change | 20.5 (15) | 14.8 (10.9)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.17, t-test, 2 sided

4. Secondary Outcome: Measurement of Change in Kyphotic (Cobb) Angle Following Kyphoplasty
Description: Preoperative and postoperative thoracolumbar radiographs used to calculate the change in kyphotic (Cobb) angle of the spine following surgery
Time Frame: Preoperative assessment within 3 weeks before surgery and postoperative day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 14 | 17
percent change | 4.80 (4.0) | 4.70 (4.6)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.93, t-test, 2 sided

5. Secondary Outcome: Comparison of 3 Month RDQ Score Between Unipedicular and Bipedicular Kyphoplasty Groups
Description: as for outcome 2
Time Frame: 3 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Unipedicular Kyphoplasty: Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm only vertebral body pedicle was entered to deliver bone cement.
  A guidewire was placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated until the balloon was in contact with the subchondral plate, lateral vertebral body wall, or anterior cortex of the vertebral body. The balloon was then deflated and removed. Subsequently, cement was injected into the cavity and allowed to harden.
- Bipedicular Kyphoplasty Group: Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm two pedicles were entered to deliver bone cement.
  A guidewire was then placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated until the balloon was in contact with the subchondral plate, lateral vertebral body wall, or anterior cortex of the vertebral body. The balloon was then deflated and removed. Subsequently, cement was injected into the cavity and allowed to harden.
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 18 | 18
units on a scale | 11.2 (2.3) | 8.1 (3.4)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.17, t-test, 2 sided

6. Secondary Outcome: Comparison of 3 Month VAS Score Between Unipedicular and Bipedicular Kyphoplasty Groups
Description: A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.[1] It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. The scale is from 1-10 with 10 as the highest level of pain, and 0 being no pain
Time Frame: 3 months post-op
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Unipedicular Kyphoplasty: Balloon kyphoplasty achieves reduction of the vertebral compression fracture using a balloon tamp inserted into the vertebral body by a transpedicular approach, followed by fixation of the fracture fragments with polymethylmethacrylate (PMMA) bone cement. In this arm only vertebral body pedicle was entered to deliver bone cement.
  A guidewire was then placed through the Jamshidi needle, and the needle removed. A series of dilating cannulae were then advanced over the guidewire until a working cannula was in place. A 15 millimeter (mm) or 20 mm bone tamp (Kyphon Inc; Sunnydale, CA) was then introduced into the vertebral body via the cannula and inflated until the balloon was in contact with the subchondral plate, lateral vertebral body wall, or anterior cortex of the vertebral body. The balloon was then deflated and removed. Subsequently, cement was injected into the cavity and allowed to harden.
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 18 | 18
units on a scale | 4.3 (2.6) | 3.9 (2.8)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.67, t-test, 2 sided

7. Secondary Outcome: Comparison of 12 Month ODI Score Between Unipedicular and Bipedicular Kyphoplasty Groups
Description: Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.[2] The scores for all questions answered are summed. Zero is equated with no disability and 50 is the maximum disability possible
Time Frame: 12 months post-op
Population: From the period of intervention to 12 month follow-up, 9 total patients were lost in the unipedicular kyphoplasty arm, resulting in analysis of 14 patients from this arm at 12 months. 6 total patients were lost in the bipedicular kyphoplasty arm, resulting in analysis of 15 patients from this arm at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 14 | 15
units on a scale | 14.8 (10.2) | 14.1 (9.3)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.90, t-test, 2 sided

8. Secondary Outcome: Comparison of 12 Month RDQ Score Between Unipedicular and Bipedicular Kyphoplasty Groups
Description: The Roland Morris Disability Questionnaire is a widely used health status measure for low back pain. The RMDQ is scored by adding up the number of items checked by the patient. The score can therefore vary from 0 to 24. It is not recommended to give patients a 'Yes' / 'No' option. If patients indicate in any way that an item is not applicable to them, the item is scored 'No', i.e. the denominator remains 24. A score of 0 indicates no back pain, while a score of 24 indicates significant back pain.
Time Frame: 12 months post-op
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 14 | 15
units on a scale | 8.1 (11.2) | 6.7 (9.4)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.36, t-test, 2 sided

9. Secondary Outcome: Comparison of 12 Month VAS Score Between Unipedicular and Bipedicular Kyphoplasty Groups
Description: as for outcome 6
Time Frame: 12 months post-op
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 14 | 15
units on a scale | 3.7 (1.9) | 3.5 (2.0)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.87, t-test, 2 sided

10. Secondary Outcome: Middle Vertebral Body Height Restoration Following Surgery With Kyphoplasty
Description: Preoperative and postoperative thoracolumbar radiographs were used to calculate the percent changes of the middle vertebral body heights.
Time Frame: Preoperative assessment within 3 weeks before surgery and postoperative day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Number analyzed (Participants) | 14 | 17
percent change | 17.8 (12.8) | 13.7 (8.9)
Statistical Analysis 1: Comparison: Unipedicular Kyphoplasty vs Bipedicular Kyphoplasty Group; Test type: Superiority; p = 0.24, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Unipedicular Kyphoplasty | Bipedicular Kyphoplasty Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/44
Other Adverse Events (participants affected / at risk) | 0/40 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No